CLINICAL TRIAL: NCT05187104
Title: Treatment of Age-related Macular Degeneration Using Retinal Stem and Progenitor Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_Retinal
Record Dates: First submitted 2021-12-24; First posted 2022-01-11 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with age-related macular degeneration receiving standard treatment and retinal stem cells (Experimental): Patients with age-related macular degeneration receiving standard treatment and autologous retinal stem and progenitor cells
  Interventions: Biological: Cultured retinal stem and progenitor cells; Other: Standard treatment according to the clinical protocols
- Patients with age-related macular degeneration receiving standard treatment (Active Comparator): Patients with age-related macular degeneration receiving standard treatment
  Interventions: Other: Standard treatment according to the clinical protocols

INTERVENTIONS:
Biological: Cultured retinal stem and progenitor cells — Cultured retinal stem and progenitor cells injected subretinally
  Arms: Patients with age-related macular degeneration receiving standard treatment and retinal stem cells
Other: Standard treatment according to the clinical protocols — Standard treatment of age-related macular degeneration according to the clinical protocols

SUMMARY:
Treatment of age-related macular degeneration using retinal stem and progenitor cells

DETAILED DESCRIPTION:
The aim of the project is to develop a biomedical cell product based on retinal pigment epithelium cells for highly effective treatment age-related macular degeneration; to conduct the clinical trials of the biomedical cell product in the treatment of age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of age-related macular degeneration
* The patient can read, understand, follow the examination procedures and complete, if necessary, the required documentation
* Written informed consent

Exclusion Criteria:

* The presence of any malignant tumor within the last 5 years
* Acute or chronic diseases in the stage of decompensation
* Chronic infectious diseases: HIV, viral hepatitis B, C, tuberculosis
* Patients who are pregnant, breastfeeding, or fertile patients who are not using adequate contraceptive methods
* Chronic and protracted mental disorders, all diseases with the presence of the syndrome of dependence on alcohol, drugs and psychoactive substances, any other condition that makes the patient unable to understand the nature, extent and possible consequences of the study or, in the opinion of the researcher, prevents the patient from observing and performing protocol
* Patients are unable or unwilling to give written informed consent and / or follow research procedures
* Any other medical condition that, in the opinion of the investigator, may be associated with an increased risk to the patient or may affect the outcome or evaluation of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 month
  Determination of visual acuity after the therapy
Visual acuity | 1 year
  Determination of visual acuity after the therapy
Adverse effects associated with the therapy | 1 month
  Determination of adverse effects associated with the therapy
Adverse effects associated with the therapy | 1 year
  Determination of adverse effects associated with the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ludmila Marchenko, Prof, Study Director — Belarusian State Medical University; Zinaida Kvacheva, Dr, Study Director — the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No